CLINICAL TRIAL: NCT00878150
Title: Cognitive Behavioral Therapy for Depression After Traumatic Brain Injury
Brief Title: Life Improvement Following Traumatic Brain Injury
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jesse Fann, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40378 G; 1R21HD053736-01A1 (NIH); H133G070016 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Traumatic Brain Injury; Depression
Keywords: traumatic brain injury; TBI; head injury; brain injury; depression; major depressive disorder; cognitive behavioral therapy; CBT; counseling
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression; Craniocerebral Trauma; Brain Injuries; Depressive Disorder, Major | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telephone-based CBT (Experimental): - 12 counseling sessions over 16 weeks over the telephone
  Interventions: Behavioral: Telephone Cognitive Behavioral Therapy
- In-person CBT (Experimental): - 12 counseling sessions over 16 weeks at either Harborview Medical Center or the University of Washington Medical Center in Seattle, WA
  Interventions: Behavioral: In-person Cognitive Behavioral Therapy
- 3: Usual care (No Intervention): - No counseling sessions as part of this study, however you are free to pursue regular medical care and counseling outside of this study

INTERVENTIONS:
Behavioral: In-person Cognitive Behavioral Therapy — 12 sessions of CBT delivered in-person over 16 weeks
  Other Names: In-person CBT; Counseling; CBT
  Arms: In-person CBT
Behavioral: Telephone Cognitive Behavioral Therapy — 12 sessions of telephone-based CBT over 16 weeks
  Other Names: Telephone CBT; CBT; Counseling
  Arms: Telephone-based CBT

SUMMARY:
The purpose of this study is to test the effectiveness of a telephone-based and in-person Cognitive Behavioral Therapy (CBT) intervention for treating Major Depressive Disorder (MDD) following Traumatic Brain Injury. Participants are randomly assigned to receive one of the following: 1) Telephone-based CBT, 2) In-person CBT, or 3) Usual care (control).

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is the most prevalent psychiatric disorder in persons with traumatic brain injury (TBI) and is most common during the first several years after injury. MDD following TBI is associated with poor behavioral, health, and functional outcomes. While neurological factors contribute somewhat to the development of MDD in this population, there is evidence that numerous psychological, social and vocational factors also contribute.

There are also multiple barriers to effective treatment of MDD in persons with TBI, including:

* under-diagnosis and under-treatment 20lack of access to care due to mobility, transportation and health care benefit limitations
* TBI neurocognitive impairments
* comorbid medical and psychiatric problems, including substance abuse
* stressors such as lack of social support and work instability
* inaccurate beliefs about depression and its treatment among TBI survivors.

The investigators are conducting a three arm trial of Cognitive Behavioral Therapy (CBT) to treat Major Depression Disorder (MDD) that emerges within the first 10 years after complicated mild to severe traumatic brain injury (TBI). The overall objective of the study is to develop a 12-session telephone-based and in-person CBT program for people with TBI (CBT-TBI), and to evaluate its feasibility, acceptability, and effectiveness.

The investigators project aims are to

1. develop CBT for for Major Depression Disorder (MDD) in persons with TBI that can be delivered in-person or via the telephone
2. conduct a trial of CBT-TBI delivered either in-person or via telephone versus care as usual
3. refine the intervention and plan a definitive RCT of CBT-TBI if response rate is sufficient.

Participants are randomized to one of three groups: (1) 12 semi-weekly sessions of telephone-based CBT for depression provided by a study therapist, (2) 12 semi-weekly sessions of in-person CBT for depression provided by a study therapist, or (3) Usual Care (control). Randomization is stratified by injury severity to ensure equal proportions in each treatment group. Participants choose one of three randomization options that includes the groups to which he/she would like to be randomized:

* Option 1: Telephone counseling verses usual care
* Option 2: In-person counseling verses usual care
* Option 3: In-person counseling verses Telephone counseling verses usual care

Outcomes are assessed by a blinded research assistant at 8, 16, and 24 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for TBI within the last 10 years, and at least one month post-injury
* sustained a complicated mild to severe TBI as indicated by Glasgow Coma Scale score of 3-12 or had documented intracranial abnormalities on CT scan or had post-traumatic amnesia (PTA) of at least 7 days
* meet screening criteria for major depression
* speak English fluently
* resides in any of the the 50 United States

Exclusion Criteria:

* does not have a telephone
* does not have a stable address
* history of bipolar disorder or schizophrenia, or current psychosis or suicidal intent
* current alcohol or substance dependence (within last month)
* evidence of significant cognitive impairment on neuropsychological testing
* started on an antidepressant medication within 6 weeks or planning to start on an antidepressant within the 16-week study
* currently in psychotherapy for depression or plan to start psychotherapy for depression within the 16-week study period
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | 16 weeks, 24 weeks
Symptom Checklist-20 (SCL-20) | 16 weeks, 24 weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 16 weeks, 24 weeks
Head Injury Symptom Checklist | 16 weeks, 24 weeks
Structured Clinical Interview for DSM-IV (SCID)- Current MDD only | 16 weeks, 24 weeks
Automatic Thoughts Questionnaire | 16 weeks
Dysfunctional Attitudes Scale | 16 weeks
Environmental Reward Observation Scale (EROS) | 16 weeks
Medical Outcome Short Form- 36 (SF-36) | 16 weeks, 24 weeks
Sheehan Disability Scale | 16 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jesse R Fann, MD, MPH, Principal Investigator — University of Washington School of Medicine, Departments of Psychiatry & Behavioral Sciences and Rehabilitation Medicine; Charles H. Bombardier, PhD, Principal Investigator — University of Washington School of Medicine, Department of Rehabilitation Medicine
Locations (1):
- University of Washington School of Medicine, Seattle, Washington, United States

REFERENCES:
- [Derived] Dyer JR, Williams R, Bombardier CH, Vannoy S, Fann JR. Evaluating the Psychometric Properties of 3 Depression Measures in a Sample of Persons With Traumatic Brain Injury and Major Depressive Disorder. J Head Trauma Rehabil. 2016 May-Jun;31(3):225-32. doi: 10.1097/HTR.0000000000000177. PMID 26291629
- [Derived] Fann JR, Bombardier CH, Vannoy S, Dyer J, Ludman E, Dikmen S, Marshall K, Barber J, Temkin N. Telephone and in-person cognitive behavioral therapy for major depression after traumatic brain injury: a randomized controlled trial. J Neurotrauma. 2015 Jan 1;32(1):45-57. doi: 10.1089/neu.2014.3423. PMID 25072405
- See also: Related Info — http://www.LIFTcare.org